CLINICAL TRIAL: NCT04434625
Title: The Effect of a Predictive Model of Bowel Preparation Based on Procedure-related Factors: a Multicenter, Randomized Controlled Study
Brief Title: The Effect of a Predictive Model of Bowel Preparation Based on Procedure-related Factors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY20200614-3
Record Dates: First submitted 2020-06-14; First posted 2020-06-17 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Colonoscopy; Bowel Preparation; Predictive Model
Keywords: factors; bowel preparation; colonoscopy
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (No Intervention): Colonoscopy was performed in the control group directly.
- model-based interference group (Experimental): Patients with score ≥3 were asked to taking another dose of PEG (1.5L) within 1-2 hours. Colonoscopy was performed in afternoon (about 4h after drinking PEG). Patients with score<3 in IM group colonoscopy directly.
  Interventions: Drug: Polyethylene glycol

INTERVENTIONS:
Drug: Polyethylene glycol — Before colonoscopy, patient-related and procedure-related parameters were collected by one investigator in each center. In MI group, a procedure-based score, used for predicting inadequate bowel preparation, was calculated for each patients. Patients with score ≥3 were asked to taking another dose of PEG (1.5L) within 1-2 hours. Colonoscopy was performed in afternoon (about 4h after drinking PEG). Patients with score<3 in IM group and those in the control group underwent colonoscopy directly
  Arms: model-based interference group

SUMMARY:
The rate of adequate bowel preparation is one of important quality indicators of colonoscopy. Inadequate bowel preparation negatively affects the outcomes of colonoscopy. If patients with inadequate bowel preparation were identified before the procedure, enhanced strategy could be offered to achieve better bowel cleaning. Currently, there were three predicting models of inadequate bowel preparation established based on patient-related factors. So far, none of predictive models have been tested in other than their validation cohort populations, and no study has attempted to apply a different regimen to patients presenting with risk factors for inadequate colon cleanliness. In previous studies, we established a prediction model based on procedure-related factors, which has better accuracy and can better predict the quality of bowel preparation.

The aim of this study is to compare the quality of bowel preparation by using a predictive model based on procedure-related factors versus the criterion group in unsedation patients

ELIGIBILITY:
Inclusion Criteria:

* Age: 18~75 years
* Patients undergoing morning colonoscopy

Exclusion Criteria:

* colon resection;
* suspected bowel obstruction;
* moderate or severe complications related to drinking the 1st or 2rd dose of PEG
* hemodynamically unstable;
* lactating or pregnant women;
* no need to reach the ileocecal segment
* unwilling to provided informed content.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 900 (Actual)
Dates: Start 2020-06-14 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation | 6 months
  Defined by each segmental BBPS≥2

SECONDARY OUTCOMES:
Adenoma detection rate | 6 months
  The proportion of participants with at least one adenoma in each group
Overall complication related to bowel preparation | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, M.D, Study Chair — Air Force Military Medical University, China
Locations (5):
- China (5):
  - Department of Gastroenterology, Hongai Hospital, Xiamen, Fujian
  - Department of Holistic Integrative Medicine, Shenzhen Hospital of Southern Medical University, Shenzhen, Guangdong
  - Department of Gastroenterology, Huaihe Hospital of Henan University, Kaifeng, Henan
  - Department of Gastroenterology, Shaanxi Second People's Hospital, Xi'an, Shaanxi
  - Endoscopic center, Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi

REFERENCES:
- [Background] Hassan C, Fuccio L, Bruno M, Pagano N, Spada C, Carrara S, Giordanino C, Rondonotti E, Curcio G, Dulbecco P, Fabbri C, Della Casa D, Maiero S, Simone A, Iacopini F, Feliciangeli G, Manes G, Rinaldi A, Zullo A, Rogai F, Repici A. A predictive model identifies patients most likely to have inadequate bowel preparation for colonoscopy. Clin Gastroenterol Hepatol. 2012 May;10(5):501-6. doi: 10.1016/j.cgh.2011.12.037. Epub 2012 Jan 10. PMID 22239959
- [Background] Dik VK, Moons LM, Huyuk M, van der Schaar P, de Vos Tot Nederveen Cappel WH, Ter Borg PC, Meijssen MA, Ouwendijk RJ, Le Fevre DM, Stouten M, van der Galien O, Hiemstra TJ, Monkelbaan JF, van Oijen MG, Siersema PD; Colonoscopy Quality Initiative. Predicting inadequate bowel preparation for colonoscopy in participants receiving split-dose bowel preparation: development and validation of a prediction score. Gastrointest Endosc. 2015 Mar;81(3):665-72. doi: 10.1016/j.gie.2014.09.066. Epub 2015 Jan 17. PMID 25600879
- [Background] Gimeno-Garcia AZ, Baute JL, Hernandez G, Morales D, Gonzalez-Perez CD, Nicolas-Perez D, Alarcon-Fernandez O, Jimenez A, Hernandez-Guerra M, Romero R, Alonso I, Gonzalez Y, Adrian Z, Carrillo M, Ramos L, Quintero E. Risk factors for inadequate bowel preparation: a validated predictive score. Endoscopy. 2017 Jun;49(6):536-543. doi: 10.1055/s-0043-101683. Epub 2017 Mar 10. PMID 28282690
- [Derived] Chen L, Kang X, Ren G, Luo H, Zhang L, Wang L, Zhao J, Zhang R, Zhang X, Zhao L, Pan Y. Individualized intervention based on a preparation-related prediction model improves adequacy of bowel preparation: A prospective, multi-center, randomized, controlled study. Dig Liver Dis. 2024 Mar;56(3):436-443. doi: 10.1016/j.dld.2023.09.001. Epub 2023 Sep 19. PMID 37735023